CLINICAL TRIAL: NCT02194634
Title: Safety and Efficacy Study of Conbercept in Diabetic Macular Edema (DME) (Sailing)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KHSWKH902010
Record Dates: First submitted 2014-07-14; First posted 2014-07-18 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-06

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — KH902 fusion protein; salicylhydroxamic acid; Lasers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conbercept treatment group (Experimental): Conbercept injection and sham laser treatment at day 0 for 1st time, the investigators will decide whether the subjects need to get repeated treatment according to monthly assessment.
  Interventions: Drug: Conbercept; Other: Sham laser
- Laser treatment group (Active Comparator): Laser treatment and sham injection at day 0 for 1st time, the investigators will decide whether the repeated laser treatment is needed according to monthly results during the visit after 3 months.
  Interventions: Other: Sham injection; Procedure: Laser

INTERVENTIONS:
Drug: Conbercept — Intravitreal injection of 0.5 mg Conbercept at first month, then repeated as needed.
  Arms: Conbercept treatment group
Other: Sham injection — Sham intravitreal injection at first month, then repeated as needed.
  Arms: Laser treatment group
Procedure: Laser — Laser treatment at first month, then repeated as needed.
  Arms: Laser treatment group
Other: Sham laser — Sham laser at first month, then repeated as needed.
  Arms: Conbercept treatment group

SUMMARY:
This study is designed to assess safety and efficacy of intravitreal injection of Conbercept on visual acuity and anatomic outcomes in patients with diabetic macular edema (DME) .

ELIGIBILITY:
Inclusion Criteria:

1. Patients sign informed consent, and are willing and able to comply with all the follow-ups;
2. Age ≥ 18 years , both genders;
3. Diagnosis of type 1 or type 2 diabetes mellitus;
4. Serum HbA1c ≤ 10%;
5. Study eye must meet the following criteria:

   * Visual acuity impairment caused by DME with involving foveal;
   * BCVA score ≥ 24 and ≤ 73 Early Treatment Diabetic Retinopathy Study (ETDRS) letters at 4 meter/1 meter of ETDRS test(Equivalent Snellen chart 20/40 to 20/320);
   * Visual impairment due to Choroidal Neovascularization (CNV) secondary to high myopia.
   * Central retinal thickness (CRT) ≥300μm (spectral domain Optical Coherence Tomography (OCT), the CRT measurements must be confirmed by central reading center);
   * Refractive media opacities and miosis have no effect on the fundus examination.
6. Non-study eye BCVA ≥ 24 letters (equivalent to Snellen visual acuity 20/320).

Exclusion Criteria:

1. Active infectious ocular inflammation in either eye;
2. Proliferative diabetic retinopathy (PDR) in the study eye, with the exception of inactive, regressed PDR;
3. Any other ocular disorder in the study eye that may cause macular edema excluded the diabetic retinopathy;
4. Iris neovascularization in the study eye;
5. Uncontrolled glaucoma, or history of glaucoma surgery;
6. Aphakia in the study eye;
7. History of vitrectomy in the study eye;
8. History of panretinal laser photocoagulation (PRP) in the study eye 6 months prior to the screening, or possibly need panretinal photocoagulation of the study eye during the study;
9. Liver, kidney dysfunction;
10. History of allergic reaction to fluorescein, protein agents for diagnosis or therapy, or more than 2 drug or nondrug factors, or concomitant allergic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in best corrected visual acuity (BCVA) at month 12 | Baseline and month 12
  To compare mean change from baseline BCVA between treatment group and controlled group at month 12.

SECONDARY OUTCOMES:
Mean change from baseline in central retinal thickness (CRT) between two groups | Baseline and month 12
  To compare mean change from baseline CRT between two groups at month 12.
Safety (e.g. incidence of adverse events) of Conbercept ophthalmic injection | 12 months
  To assess safety parameters during the study, such as incidence of adverse events , incidence of adverse drug reactions etc.

OTHER OUTCOMES:
Mean changes from baseline of photographic parameters, such as CRT, total macular volume and leakage area etc. | Baseline and every month, up to 12 months
Mean change from baseline BCVA between treatment group and controlled group | Baseline and every month, up to 12 months
Change from baseline in visual acuity distribution of treatment group and controlled group | Month 6, month 12
The 25-item National Eye Institute Visual Function Questionnaire （NEI VFQ-25）total score mean change from baseline of between treatment group and controlled group | Month 6, month 12

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tongren hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Daping Hospital, Research Institute of Surgery Third Military Medical University, Chongqing, Chongqing Municipality
  - Zhongshan Ophthalmic Center , Sun Yat-Sen University, Guangzhou, Guangdong
  - Eye hospital of Henan province, Zhengzhou, Henan
  - Wuhan General Hospital of Guangzhou Military, Wuhan, Hubei
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - He eye hospital, Shenyang, Liaoning
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Renji hospital shanghai jiaotong university school of medcine, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xian, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Eye center of Tianjin mendical university, Tianjin, Tianjin Municipality
  - The Affiliated Eye Hospital of WMC, Wenzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing

REFERENCES:
- [Derived] Liu K, Wang H, He W, Ye J, Song Y, Wang Y, Liu X, Wu Z, Chen S, Fan K, Liu Y, Zhang F, Li Z, Liu L, Zhang J, Zhang X, Ye J, Liang X, Li X, Ke X, Wu Q, Li J, Tao S, Wang X, Rosenfeld P, Heier JS, Kaiser P, Xu X. Intravitreal conbercept for diabetic macular oedema: 2-year results from a randomised controlled trial and open-label extension study. Br J Ophthalmol. 2022 Oct;106(10):1436-1443. doi: 10.1136/bjophthalmol-2020-318690. Epub 2021 May 17. PMID 34001667